CLINICAL TRIAL: NCT02094534
Title: A Prospective, Randomized, Double-blind, Placebo Controlled Study to Assess the Impact of ORMD-0801 (Insulin Capsules) on the Exogenous Insulin Requirements of Type 1 Diabetics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oramed, Ltd. (Industry)
Collaborators: Integrium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ORA-D-010
Record Dates: First submitted 2014-03-20; First posted 2014-03-24 (Estimated); Results first posted 2017-07-06 (Actual); Last update posted 2017-07-06 (Actual); Status verified 2017-06

CONDITIONS: Diabetes Mellitus Type 1
Keywords: Diabetes type 1; Oral Insulin; Safety; Tolerability; Phase 2a; Randomized; Blinded; Parallel
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — ORMD-0801; Insulin; Fish Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ORMD-0801 Capsules (Experimental): API (recombinant human insulin USP), in Oramed's proprietary formulation in capsules, ORMD-0801
  Interventions: Biological: ORMD-0801 Capsules
- Placebo (Placebo Comparator): Fish oil in capsules, identical in appearance to ORMD-0801
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: ORMD-0801 Capsules — API (recombinant human insulin USP), in Oramed's proprietary formulation in capsules.
  Other Names: Oral Insulin
  Arms: ORMD-0801 Capsules
Other: Placebo — Fish oil capsules, identical in appearance to the experimental intervention.
  Other Names: Fish Oil
  Arms: Placebo

SUMMARY:
This will be a prospective, randomized, double-blind, placebo controlled study. Patients with established Type 1 diabetes will be eligible for entry into the study. Eligible patients will be screened and those who fulfill all inclusion/exclusion criteria will be admitted to the inpatient unit no fewer than 2 days and no more than 7 days after Screening. Patients will report to the inpatient unit at 6 a.m. and outfitted with a continuous glucose monitoring (CGM) device. Patients will be given standardized meals and snacks for the duration of their inpatient visit.

DETAILED DESCRIPTION:
For the first 3 days, patients will be dosed with placebo 45 minutes prior to each of the day's 3 meals to establish baseline insulin requirements. Patients will be dosed with exogenous insulin according to their normal sliding scale and each patient's daily insulin requirement will be documented. The average daily insulin requirements during the 3 day run-in period will constitute the patient's baseline insulin level.

Following the 3 day run-in, the CGM device will be detached, its data download, and the patient refitted with the CGM with a fresh cannula for continued monitoring during the 7-day treatment period.

Patients will be randomized 2:1 to receive ORMD-0801 or placebo for the 7-day double-blind treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females age 18 to 55 years old, inclusive.
* Patients must be willing and able to sign informed consent.
* Documented history of Type 1 Diabetes for at least 6 months
* Females of childbearing potential must have a negative serum pregnancy test at screening and a negative urinary screening test following admission to the inpatient unit

Exclusion Criteria:

* Presence of any clinically significant endocrine disease according to the Investigator (euthyroid patients on replacement therapy will be included if the dosage of thyroxine is stable for at least six weeks prior to Screening)
* Fasting plasma glucose >260 mg/dL at the end of run-in
* Evidence of unawareness of hypoglycemia with a documented plasma glucose ≤50 mg/dL in the absence of symptoms of hypoglycemia
* Presence of any clinically significant condition that might interfere with the evaluation of study medication (i.e., significant renal, hepatic, gastrointestinal (GI), cardiovascular (CV), immune disease).
* Presence or history of cancer within the past five years with the exception of adequately-treated localized basal cell skin cancer or in situ uterine cervical cancer
* Laboratory abnormalities at screening including:
* Positive pregnancy test in females of childbearing potential (at screening and Day -3 of Visit 2)
* Abnormal serum thyrotropin (TSH) levels >1.5X upper limit of normal (ULN)
* Positive test for hepatitis B surface antigen and/or hepatitis C antibody
* Positive test for HIV
* Any relevant abnormality interfering with the efficacy or the safety assessments during study drug administration
* Use of the following medications:

  o History of use of aprotinin at any time prior to the screening visit (e.g., Trasylol, any type or dose)
* Administration of thiazolidinedione [e.g., (Actos (pioglitazone) and Avandia (rosiglitazone)] treatment within 3 months prior to randomization.
* Administration of thyroid preparations or thyroxine (except in patients on stable replacement therapy) within 6 weeks prior to screening visit
* Administration of systemic long-acting corticosteroids within two months or prolonged use (more than one week) of other systemic corticosteroids or inhaled corticosteroids (if daily dosage is > 1,000 μg equivalent beclomethasone) within 30 days prior to screening visit
* Use of medications known to modify glucose metabolism or to decrease the ability to recover from hypoglycemia such as oral, parenteral, and inhaled steroids (as discussed above), beta blockers (with the exception of beta blocker ophthalmic solutions for glaucoma or ocular hypertension), and immunosuppressive or immunomodulating agents
* History of severe or multiple allergies, or known allergy to soy or aprotinin.
* History of tobacco or nicotine use within 10 weeks prior to screening
* Patient is on a weight loss program and is not in the maintenance phase, or patient that started weight loss medication (e.g., orlistat or sibutramine) within 8 weeks prior to screening
* Pregnancy or breast-feeding
* Patient has a screening visit systolic blood pressure of ≥165 mmHg or diastolic blood pressure of ≥100 mmHg.
* Patient is, at the time of consent, a user of recreational or illicit drugs or has had a recent history (within the last year) of drug or alcohol abuse or dependence. (Note: Alcohol abuse includes heavy alcohol intake as defined by >3 drinks per day or >14 drinks per week, or binge drinking)
* Elevated liver enzymes (alanine transaminase (ALT), alanine aminotransferase (AST), alkaline phosphatase) greater than 2 times the upper limit of normal (ULN) at Screening
* Very high triglyceride level (>600 mg/dL) at Screening
* Any clinically significant electrocardiogram (ECG) abnormality at screening or cardiovascular disease. Clinically significant cardiovascular disease will include:
* history of stroke, transient ischemic attack, or myocardial infarction within 6 months prior to screening,
* history of or currently have New York Heart Associate Class II-IV heart failure prior to screening, or
* uncontrolled hypertension defined as (duplicate seated reading) blood pressure ≥165 mmHg (systolic) or ≥100 mmHg (diastolic) at screening or at Visit 2.
* History of gastrointestinal disorders (e.g. hypochlorhydria) with the potential to interfere with drug absorption
* At the Principal Investigator's discretion, any condition or other factor that is deemed unsuitable for patient enrollment into the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2014-03; Primary Completion 2014-08 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Kidron, Ph.D., Study Director — Oramed, Ltd.
Locations (1):
- Orange County Research Center, Tustin, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects took all doses of intervention.
Pre-assignment Details: Basal Exogenous Insulin - Intend to Treat (ITT) - All Subjects
Groups:
- ORMD-0801: API (recombinant human insulin USP), in Oramed's proprietary formulation in capsules, ORMD-0801
  ORMD-0801 capsules: API (recombinant human insulin USP), in Oramed's proprietary formulation in capsules.
Period: Overall Study
Arm/Group | ORMD-0801 | Placebo
Started | 15 | 10
Completed | 15 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ORMD-0801 | Placebo | Total
Number analyzed (Participants) | 15 | 10 | 25
Age, Categorical [Count of Participants; unit: Participants] — 3 Day Placebo Run-in Period
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 15 | 10 | 25
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.90 (11.936) | 37.61 (9.642) | 38.255 (15.343)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 12 | 5 | 17
Region of Enrollment [Number; unit: participants]
  United States | 15 | 10 | 25

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total, Basal, and Bolus Exogenous Insulin Requirements
Description: Change from baseline (Run-in Average) to treatment days 6 and 7 (average of day 6 and 7) in exogenous insulin requirements in patients treated with ORMD-0801 compared to patients treated with placebo.
Time Frame: Baseline:Run-In Average (run in days 1-7), and treatment (day 6 and day 7)
Population: Intend-to-treat polpulation
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | ORMD-0801 | Placebo
Number analyzed (Participants) | 15 | 10
mg/dL
  Total Exogenous Insulin Usage | -2.09 (10.936) | 2.83 (12.716)
  Basal Exogenous Insulin Usage | -1.92 (7.517) | -1.10 (10.423)
  Bolus Exogenous Insulin Usage | -0.18 (10.310) | 3.93 (6.541)

2. Secondary Outcome: Mean Nighttime, Daytime, and Fasting Glucose Levels
Description: Mean glucose levels (by continuous glucose monitoring (CGM)) in Type 1 diabetes patients treated with ORMD-0801, compared to the mean glucose levels (by continuous glucose monitoring) for patients treated with placebo.
Time Frame: last two days (day 6 and day 7, averaged)
Population: Intent to treat (ITT) population; This measurement is reported for those subjects who had at least 80% of the CGM readings. This explains why there are two fewer subjects from the ITT population reported for this endpoint.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | ORMD-0801 | Placebo
Number analyzed (Participants) | 14 | 9
mg/dL
  Mean nighttime levels by CGM | 137.65 (31.311) | 133.17 (23.321)
  Mean daytime glucose levels by CGM | 145.15 (18.408) | 165.73 (19.372)
  Mean fasting glucose levels by CGM | 122.15 (32.670) | 138.69 (35.295)

ADVERSE EVENTS:
Time Frame: Three Months
Description: Adverse Events of Hypoglycemia The CTCAE (version 4.0) definition for mild, moderate, and severe hypoglycemia based on blood glucose will be used, as shown below: Mild: from 55 to <70 mg/dL Moderate: from 40 to < 55 mg/dL Severe: from 30 to < 40 mg/dL Life Threatening: < 30 mg/dL (< 1.7 mmol/L)
Arm/Group | ORMD-0801 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/10
Other Adverse Events (participants affected / at risk) | 15/15 | 10/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ORMD-0801 (N=15) | Placebo (N=10)
Hypoglycemia (Metabolism and nutrition disorders) | 15 (201) | 10 (124)
Hyperglycemia (Metabolism and nutrition disorders) | 13 (51) | 9 (41)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) — Treatment-Emergent Adverse Events by System Organ Class, and Preferred Term
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — Treatment-Emergent Adverse Events by System Organ Class, and Preferred Term
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Treatment-Emergent Adverse Events by System Organ Class, and Preferred Term
Fatigue (General disorders) | 1 (1) | 0 (0) — Treatment-Emergent Adverse Events by System Organ Class, and Preferred Term
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Treatment-Emergent Adverse Events by System Organ Class, and Preferred Term
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Treatment-Emergent Adverse Events by System Organ Class, and Preferred Term
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) — Treatment-Emergent Adverse Events by System Organ Class, and Preferred Term
Head discomfort (Nervous system disorders) | 1 (1) | 0 (0) — Treatment-Emergent Adverse Events by System Organ Class, and Preferred Term
Headache (Nervous system disorders) | 2 (2) | 1 (1) — Treatment-Emergent Adverse Events by System Organ Class, and Preferred Term
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Treatment-Emergent Adverse Events by System Organ Class, and Preferred Term

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Agreement is "work for hire"